CLINICAL TRIAL: NCT05450887
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Obeticholic Acid in Patients With Primary Biliary Cholangitis
Brief Title: Efficacy and Safety of Obeticholic Acid in the Treatment of Primary Biliary Cholangitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABDSP2021-III
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCA 5 mg titrated to 10 mg ± UDCA (Experimental): OCA 5 mg once daily for 3 months and then titrating up to 10 mg based on tolerability and response.
  Subjects receiving UDCA continued taking UDCA throughout the trial. If the subjects could not tolerate UDCA, they were not treated with UDCA.
  Interventions: Drug: Obeticholic Acid Tablets（OCA）; Drug: UDCA
- Placebo ± UDCA (Placebo Comparator): Placebo once daily. Subjects receiving UDCA continued taking UDCA throughout the trial. If the subjects could not tolerate UDCA, they were not treated with UDCA.
  Interventions: Drug: UDCA; Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid Tablets（OCA） — Obeticholic Acid：Once a day (QD) by mouth (PO).
  Arms: OCA 5 mg titrated to 10 mg ± UDCA
Drug: UDCA — UDCA：13~15 mg/kg/day
Drug: Placebo — Placebo：Once a day (QD) by mouth (PO).
  Arms: Placebo ± UDCA

SUMMARY:
Obecholic acid is a modified bile acid and Farnesoid X receptor (FXR) agonist. FXR is a key regulator of bile acid synthesis and transport. Bile acids are used by the body to help with digestion. Conventional therapy with obecholic acid will improve liver function of patients with (primary biliary cholangitis)PBC.

The main objectives of the study were to assess the effects of Obeticholic Acid (OCA) on serum alkaline phosphatase (ALP) and total bilirubin, together as a composite endpoint and on safety in participants with PBC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years；
2. Definite PBC diagnosis, as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors: ① Indicators reflecting cholestasis such as elevated ALP；② Positive antimitochondrial antibody (AMA) or AMA-M2, or positive PBC-specific antibody (anti-GP210 and/or anti-SP100) if AMA negative；③ Liver biopsy consistent with PBC；
3. At least 1 of the following qualifying biochemistry values: ① ALP ≥ 1.67x ULN ；② Total bilirubin > ULN but < 2x ULN；
4. Taking UDCA for at least 6 months (stable dose for ≥ 3 months) prior to Day 0, or unable to tolerate UDCA (no UDCA for ≥ 3 months) prior to Day 0；
5. Understand the study, comply with the study protocol, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients who took obeticholic acid within 3 months prior to Day 0;
2. Known hypersensitivity to obeticholic acid, ursodeoxycholic acid;
3. History or presence of other concomitant liver diseases;
4. Cirrhosis-related complications or end-stage liver disease manifestations;
5. Serum creatinine (Cr) ≥ 1.5 × ULN and serum creatinine clearance < 60 mL/min;
6. Patients with severe pruritus or requiring systemic drug therapy within 2 months prior to Day 0;
7. Patients with HIV or syphilis infection;
8. Presence of diseases or physiological conditions that interfere with the absorption, distribution, metabolism or excretion of test drugs, such as inflammatory bowel disease and previous gastric bypass surgery;
9. Presence of diseases that may cause non-hepatogenic ALP elevation, or diseases that may lead to a life expectancy of less than 2 years;
10. Administration of the following drugs within 6 months prior to Day 0: azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, pentoxifylline; fenofibrate or other fibrates; budesonide and other systemic corticosteroids; hepatotoxic drugs (including α-methyldopa, sodium valproate, isoniazid, nitrofurantoin, etc.);
11. Administration of the following drugs within 12 months prior to Day 0: antibodies or immunotherapy against interleukins or other cytokines or chemokines;
12. Patients with serious cardiovascular system, digestive system, respiratory system, urinary system, nervous system, mental illness, immunodeficiency disease, and judge by investigators that they are not suitable for participating in the trial;
13. Other conditions that are not considered appropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Percentage of PBC patients reaching the compound endpoint after 12 months of treatment (Compound endpoint: alkaline phosphatase (ALP) < 1.67× Upper Limit of Normal(ULN), and ALP decrease ≥ 15% from baseline, and total bilirubin ≤ ULN ) | up to 12 months
  Compound endpoint: ALP < 1.67× ULN, and ALP decrease ≥ 15% from baseline, and total bilirubin ≤ ULN

SECONDARY OUTCOMES:
Absolute change and percentage change of ALP, total bilirubin, direct bilirubin, ALT, AST and GGT from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for ALP, total bilirubin, direct bilirubin, ALT, AST and GGT levels. Absolute change and percentage change of ALP, total bilirubin, direct bilirubin, ALT, AST and GGT from baseline to Month 3, 6, 9 and 12 are presented.
Quality of life for PBC measure (PBC-40) score percentage change from baseline to Month 3, 6, 9 and 12 | up to 12 months
  PBC-40 score was evaluated at certain visits. PBC-40 score percentage change from baseline to Month 3, 6, 9 and 12 is presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China